CLINICAL TRIAL: NCT01606813
Title: The Impact of Integrating an Internet Weight Control Program Into Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of North Carolina, Chapel Hill (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor; Division Chief of General Internal Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 39237EP; 1R01DK095078-01 (NIH)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief physician counseling (BPC) + Usual care (UC) (Active Comparator): The participant will receive standard care. They will receive BPC from their PCP on weight loss by reviewing a goal setting worksheet and collaboratively setting a goal for weight loss.
  Interventions: Other: Usual Care; Behavioral: Brief Physician Counseling
- BPC + Internet Weight Control Program (IWCP) (Experimental): The participant will receive BPC from their PCP by reviewing a goal setting worksheet and collaboratively setting a goal for weight loss. They will receive referral and access to an internet weight control program.
  Interventions: Behavioral: Brief Physician Counseling; Behavioral: Referral and access to an internet weight control program
- BPC + IWCP + Follow up email notes from PCP (Experimental): The participant will receive BPC form their PCP by reviewing a goal setting worksheet and collaboratively setting a goal for weight loss. They will receive referral and access to an internet weight control program. And they will receive brief follow up email notes from PCPs on how their weight loss is going (from data collected from the weight loss website).
  Interventions: Behavioral: Brief Physician Counseling; Behavioral: Referral and access to an internet weight control program; Behavioral: Brief follow up email notes from PCPs

INTERVENTIONS:
Other: Usual Care — Standard care
  Arms: Brief physician counseling (BPC) + Usual care (UC)
Behavioral: Brief Physician Counseling — Primary Care Physician (PCP) will review a goal setting worksheet for weight loss with the participant and then collaboratively set a goal for weight loss.
Behavioral: Referral and access to an internet weight control program — Participants will receive a login and password for the weight loss website. The website will encourage patients to set a new weight goal every 3 months and work towards a total weight loss goal of 10%. Patients will also receive an email prompt each week alerting them to new content and reminding them to check-in to the website to report their weight, intake and activity.
  Arms: BPC + IWCP + Follow up email notes from PCP; BPC + Internet Weight Control Program (IWCP)
Behavioral: Brief follow up email notes from PCPs — Patients will receive a biweekly email from their primary care physician on how they are doing with their weight loss.
  Arms: BPC + IWCP + Follow up email notes from PCP

SUMMARY:
The investigators will conduct a randomized controlled trial comparing the effects of three interventions on weight loss at 12 months. The investigators propose to test the impact of integrating an effective automated Internet weight control program into primary care by recruiting patients and randomizing them to one of three conditions: A) Brief physician counseling plus usual care, B) Brief physician counseling plus referral and access to the Internet weight control program and, C) Brief physician counseling plus referral and access to the Internet weight control program plus brief follow-up email notes of support and accountability from Primary Care Physicians. The investigators hypothesize that an online program for weight control can be more effective by enhancing online follow-up with PCPs.

DETAILED DESCRIPTION:
Every year, roughly 700 of the 750 million visits that overweight and obese patients make with primary care providers (PCPs) occur without any weight counseling. The main reasons for this are that PCPs are poorly trained to help their patients lose weight and that there are no consistently effective interventions for primary care settings. Though in-person and telephone-based weight control programs have been difficult to disseminate in primary care, online weight control programs are increasingly effective and may lend themselves to be used in these settings. Given the growing number of effective online programs, for obesity and for other conditions seen in primary care (e.g., depression, insomnia) it is important to understand whether these programs can be effective when integrated into primary care and whether they are enhanced by provider involvement. Research on the 5 A's model of primary care behavior change suggests that the most effective, yet least used feature of primary care interventions is arranging follow-up, where providers hold patients accountable to adhering to treatments and achieving specific outcomes.

The 5 A's model provides a useful framework for integrating behavior change interventions into primary care. In this model, providers ASK about weight, ADVISE patients to lose weight, ASSESS readiness to change, ASSIST the patient in making changes and ARRANGE follow-up. Unfortunately, though PCPs are uniquely positioned to ARRANGE follow-up, given their long-term relationship with the patient, and studies show that ARRANGING follow-up may be the most effective of the 5 A's, it is the least often used. In a study of 481 encounters with overweight patients, Pollak (Consultant) and colleagues observed that PCPs ARRANGED follow-up in only 5% of visits, though it was the only one of the 5 A's associated with future weight loss. Kottke and colleagues similarly observed that primary care smoking cessation interventions that included more "reinforcing sessions" with PCPs were the most effective. This is consistent with conclusions by Whitlock and colleagues that "Simply notifying patients that follow-up will occur seems to be a powerful motivating factor". These findings have been extended to online interventions, where two meta-analyses concluded that the impact of online interventions for depression and anxiety is enhanced by follow-up that includes being accountable to and supported by a human being.

The investigators have created a simple method for integrating an Internet weight control program into primary care settings, by allowing PCPs to monitor their patients' adherence and outcomes and email them pre-written, tailored follow-up messages. PCPs in the investigators' pilot work believed that this would help to overcome key barriers to helping their patients lose weight.

ELIGIBILITY:
INCLUSION CRITERIA:

Physicians and Mid-level providers (Focus group and RCT):

* Has medical license to practice primary care
* Practice within 60 miles (focus group)/100 miles (RCT) of Penn State Hershey Medical Center
* Practice not located at Penn State Hershey Medical Center campus (focus group)
* Be active primary care providers (provide primary care at least 2 half days per week at one practice)
* Not have had completed a weight management fellowship
* Use internet in their office

Patients (Focus group only):

* Ages 21-60
* Body Mass Index between 25.0-50.0 kg/m2
* Have internet access at home or work
* Patient of a primary care provider who practices Internal Medicine or Family Community Medicine
* Has seen primary care provider in the last year, not including acute care

Patients (RCT only)

* Ages 21-70
* Body Mass Index between 25.0-50.0 kg/m2
* Have internet access at home or work
* Patient of a PCP who is participating in the study
* Patient has been seeing the PCP for at least 12 months and has no other PCP
* The PCP must approve the patients' participation

EXCLUSION CRITERIA:

Physicians and Mid-level providers (RCT only)

* Practice serves a specialty care population
* Pregnant or planning to become pregnant in the next 3 months
* Planning on changing practice locations in the next 12 months
* Planning on retiring in the next 12 months

Patients (Focus group and RCT)

* Losing >5% of current body weight in the previous 6 months
* Participating in a research project involving weight loss or physical activity in the previous 6 months
* Pregnancy during the previous 6 months, lactating, or planning to become pregnant in the next 3 months (focus group)/12 months (RCT)
* Planning on moving out of the area in the next 3 months (focus group)/12 months (RCT)
* Current treatment for a condition or with a medication that could impact weight (Orlistat - aka. Alli, Phentermine, Topiramate - aka. Topamax) and are not willing to stop for duration of the study
* Hospitalization for psychiatric problems during the prior year

Patients (RCT only)

* Had weight loss surgery
* Planning on changing primary care provider in the next 12 months
* Participating in an online or community weight loss program (e.g., Weight Watchers) and not willing to stop for the duration of the study
* Doctor has diagnosed a heart condition and said should only do physical activity recommended by doctor
* Feel pain in chest when doing physical activity
* In the past month, have had chest pain when not doing physical activity
* In the end stages of renal, liver or kidney diseases
* Has heart failure
* Has/had cancer in past 5 years (except non-melanoma skin cancer)
* Cannot walk for exercise for 10 minutes
* Not willing to participate in 12-month intervention
* Taking insulin
* Treated for or diagnosed with an eating disorder
* Diagnosed with HIV
* Two weeks of steroid use in past year

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 months
  Body weight and height will be measured by a research assistant using a portable, calibrated stadiometer (Tanita, Inc). Waist circumference will be measured using standard procedures, recorded to the nearest millimeter.

SECONDARY OUTCOMES:
Block Food Frequency Questionnaire | 12 months
  This questionnaire asks participants to estimate how often they consume a variety of specific foods.
Paffenbarger Activity Questionnaire | 12 months
  This instrument has been used to estimate leisure time activity in many studies of weight loss (78, 112-113) and changes in energy expenditure using this measure correlate with changes in body weight over at least an 18 month period (114). A scoring algorithm allows the calculation of caloric expenditure overall as well as in activities of light, medium and high intensity.
Patterns of medical care | 6 months
  After 12 months, data will be collected from medical charts using a standardized form to identify: 1) number of PCP visits, 2) use of any approved (e.g., Xenical) or off-label (e.g., Topiramate) weight loss medications after randomization, and 3) evaluations by a surgical weight control program.
Use of the 5 A's during PCP Visits | 12 months
  After the index PCP visit and quarterly, subjects will complete a survey detailing the use the 5 A's (Ask, Advise, Assess, Assist and Arrange) during visits. Within 24-72 hours after the index visit, subjects will be called to complete the exit interview.
Sociodemographics and tobacco use | 12 months
  Age, gender, race and ethnicity, smoking status, education and other demographics, will be measured based on standard self-report.
Weight History Questionnaire | 12 months
  To measure past weight, past weight loss attempts and methods used to lose weight in the past, we will use the Weight History Questionnaire (WHQ) from the National Health and Nutrition Examination Survey (NHANES).
Health Literacy | 12 months
  To measure health literacy, the Newest Vital Sign (NVS), a nutrition label that is accompanied by 6 questions that requires 3 minutes for administration will be used.
Three-Factor Eating Questionnaire (TFEQ) | 12 months
  The TFEQ measures three dimensions of dietary restraint: cognitive restraint, disinhibition, perceived hunger.
Depressive Symptoms | 12 months
  Depressive symptoms have been associated with body weight changes, so these symptoms will be measured with the 20-item Centers for Epidemiological Studies Depression Scale (CES-D). *If a patient scores a 25 or higher on the scale, research staff will notify their primary care physician; however, this does not make them ineligible for the study.
Treatment Self-Regulation Scale (TSRQ) | 12 months
  The TSRQ will be used to measure autonomous (5 items) versus controlled (8 items) motivations, as well as total motivation (autonomous + controlled).
Weight Control Self-Efficacy | 12 months
  Perceived competence in weight control will be measured using the Efficacy Life-Style Questionnaire (WEL). The WEL is a 20-item instrument consisting of five situational factors (Negative Emotions, Availability, Social Pressure, Physical Discomfort, and Positive Activities).
Patient Satisfaction and Accountability | 12 months
  Patient satisfaction will be measured with the Patient Satisfaction Questionnaire 18 (PSQ18), which includes scales to measure technical quality, interpersonal manner, communication and time spent with the doctor with scale reliability between 0.79 and 0.93. Accountability will be measured with a 6-item measure developed by Mohr and colleagues (consultant), which measures the extent to which subjects believe that they are being monitored and the extent to which they are concerned about being judged by the monitor.
Sedentary Behavior | 12 months
  This validated questionnaire asks participants about the duration of specific sedentary behaviors during a typical weekday and weekend day.
Physical Activity Self Efficacy | 12 months
  This questionnaire asks about participants about their level of confidence in doing physical activity in certain situations.
Eating Behavior Inventory | 12 months
  The Eating Behavior Inventory (EBI) is a validated questionnaire used by obesity researchers to measure the adoption of specific behaviors linked with weight-loss success.
Internet Usage | 12 months
  This questionnaire asks participants about the frequency of their Internet use and the ways in which they use the Internet
Analysis of text edits in PCP emails | 12 months
  We will analyze 100% of the personal notes added by PCPs to messages sent to patients in Condition C. Using a grounded theory approach, Dr. Hwang will analyze the content in the notes from PCPs and create a codebook and categories for these notes.
Blood pressure | 12 months
  Blood pressure will be measured by a research assistant using an automatic blood pressure monitor (Omron) and standard procedures.
Adherence (logins to website) | 12 months
  We will examine login data (overall and percentage of weeks logging in) as a mean and median, as well as a monthly percentage.
Medication | 12 Months
  Participants will be asked to bring their current prescription medications. The research coordinator will record the name and dose of each.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States